CLINICAL TRIAL: NCT04910607
Title: Social and Psychological Impacts of SARS-Cov-2 Pandemic Period in the Obese Population.
Acronym: OBIMPACOV
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Région Nouvelle Aquitaine (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/38
Record Dates: First submitted 2021-04-16; First posted 2021-06-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Covid19
Keywords: Obesity; COVID19; semi-directive interview
MeSH Terms: conditions — Obesity; COVID-19 | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Participating patients will be recruited from the Specialised Obesity Centres =CSO (CHU and Follow-up and rehabilitation care (SSR), as well as patient associations) to fill in a questionnaire and take part in an interview (varied panel representative of the target population in terms of place of residence, socio-professional category, sex and age).
  Interventions: Other: Questionnaire; Other: Interview
- Professional: Medical and paramedical staff involved in the partner CSOs will also be asked to participate in a semi-structured interview.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Questionnaire — Questionnaire with 4 axes:
  sociological, reflexive medical, prospective medical, transversal
  Groups: Patient
Other: Interview — Interview concerning health pathways, experience of confinement, consequences of confinement on health, representations of obesity.

SUMMARY:
The population suffering from obesity is particularly at risk during this pandemic period. The Nouvelle Aquitaine region is not spared, since according to the regional epidemiological report of 7 May 2020, carried out by Santé Publique France, 39.2% of cases admitted to the intensive care unit in Nouvelle Aquitaine and presenting risk factors are overweight or obese.

Other risk factors, such as social-environmental factors, must be taken into consideration. Socio-demographic surveys in this area highlight the socio-economic and territorial inequalities that interfere with obesity issues. Similarly, the issues of stigmatisation and isolation seem to be at the heart of the question of how to deal with these people.

DETAILED DESCRIPTION:
This is a prospective multicentre study. Participating patients will be recruited from the Specialised Obesity Centres (CHU and SSR, as well as patient associations) to fill in a questionnaire and take part in an interview (a varied panel representative of the target population in terms of place of residence, socio-professional category, sex and age).

The medical and paramedical staff involved in the partner CSOs and the patients' resources (identified by the patients' associations) will also be asked to participate in a semi-directive interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age.
* Be registered in an active file of the 3 partner CSOs.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients under protective measures or deprived of liberty:

  * pregnant or breastfeeding woman,
  * under guardianship,
  * under guardianship,
  * safeguard of justice,
  * incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The obese population is the target population of the study.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Analysed social and psychological impacts of containment | 9 months after inclusion day
  Thanks to sociology questionnaire based on the experience and paths of individuals (not a score).
  The treatments carried out will be limited to cross sorting and flat sorting, factorial analyzes and -previously- the chi-square analysis.
Consequences of social distancing during the containment | 9 months after inclusion day
  Thanks to sociology questionnaire based on the experience and paths of individuals(not a score).
  The treatments carried out will be limited to cross sorting and flat sorting, factorial analyzes and -previously- the chi-square analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud ALESSANDRIN, Dr, Study Chair — Universite de Bordeaux
Locations (3):
- France (3):
  - CHU de Limoges, Limoges
  - Hôpital Haut-Lévêque, Pessac
  - CHU de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No